CLINICAL TRIAL: NCT03245879
Title: Impact of Implementing Antibiotic Stewardship Programs in 15 Small Hospitals: A Cluster-Randomized Trial Intervention
Brief Title: Antibiotic Stewardship in Small Hospitals
Acronym: SCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Eddie Stenehjem, Associate Professor of Medicine, Intermountain Health Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1024823
Record Dates: First submitted 2017-08-03; First posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Inappropriate Prescribing; Antibiotic Stewardship; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Program 1 (Active Comparator): Implementation of a basic antibiotic stewardship program focusing on education, access to Infectious Diseases physicians, and availability of antibiotic use data.
  Interventions: Behavioral: Program 1
- Program 2 (Active Comparator): This arm increases antibiotic stewardship education and interventions. Program 2 hospitals performed audit and feedback of pre-specified antibiotics and implemented locally controlled restrictions.
  Interventions: Behavioral: Program 2
- Program 3 (Active Comparator): This arm was the most intensive antibiotic stewardship intervention. It included signficant audit and feedback, ID controlled restrictions, and ID review of designated culture/lab results.
  Interventions: Behavioral: Program 3

INTERVENTIONS:
Behavioral: Program 1 — Program 1 hospitals received a basic curriculum and tools for implementation of basic antibiotic stewardship interventions. Hospitals required an indication for every antibiotic order. A daily email was sent to a designated email account when a patient had been on an antibiotic for >48 hours. Curriculum included implementing antibiotic time-outs, IV to PO conversion, indications, evaluating for bug-drug mismatches, and recommendations on when to call the Infectious Diseases (ID) hotline. A daily antibiotic stewardship check list was created. All materials were provided to all pharmacists and remained on-site. Clinicians had access to an ID telephone hotline to answer clinical questions. Pharmacy directors and hospital leadership were provided a monthly, hospital-specific, antibiotic use dashboard. All pharmacy directors and staff received a monthly newsletter.
  Arms: Program 1
Behavioral: Program 2 — Program 2 hospitals received all the interventions of Program 1. In addition, Program 2 hospitals received more intense antibiotic stewardship education. Educational topics included audit and feedback, antibiotic de-escalation, the need for antibiotics targeting anaerobic bacteria, antibiotic allergy verification, and antibiotic restrictions. Pharmacists in Program 2 hospitals reviewed patients on vancomycin, piperacillin/tazobactam, imipenem, meropenem, and cefepime. For patients receiving one of these antibiotics, pharmacists reviewed the patients' microbiology data to identify opportunities for antibiotic de-escalation, IV to PO conversion, bug-drug mismatches, and/or indications for calling the ID hotline. Program 2 hospitals also restricted daptomycin, linezolid, imipenem, meropenem, ceftaroline, tigecycline, and all mold active antifungals. In Program 2 hospitals, the local pharmacy staff pre-authorized restricted antibiotics based on defined criteria.
  Arms: Program 2
Behavioral: Program 3 — Program 3 hospitals received all the interventions of Program 1 and Program 2. In addition, pharmacists in program 3 hospitals reviewed an expanded list of antibiotics for audit and feedback. These antibiotics included: Vancomycin, piperacillin/tazobactam, imipenem, meropenem, cefepime, ertapenem, aminoglycosides, ceftriaxone, and fluoroquinolones. Program 3 hospitals implemented the same antibiotic restrictions as Program 2 but ID pharmacists controlled pre-authorization of restricted antibiotics. In addition, an ID physician reviewed pre-specified positive cultures (e.g. all positive blood cultures, cultures with highly resistant Enterobacteraciae) and contacted providers with recommendations as needed. ID physician review occurred Monday through Friday and alerts were batched daily at 6am.
  Arms: Program 3

SUMMARY:
Core elements of effective antibiotic stewardship programs (ASPs) have been identified and evidence-based guidelines have been developed for implementation. The majority of the evidence used for these guidelines are from published studies on the effectiveness of ASPs in large academic or large community hospitals. A significant portion of healthcare in the United States, however, takes place in small hospitals. In 2015, 73% of US hospitals had < 200 beds (4,057 hospitals) and accounted for 29% of all US inpatient bed days. Limited studies on the effectiveness of antibiotic stewardship implementation have been performed in hospitals with < 200 beds. Antibiotic use rates and selection patterns in these small hospitals are similar to that of large hospitals and the majority of small hospitals lack formal ASP that meet the CDC's core elements. The objective of this real-world implementation study was to assess the effectiveness of three ASP strategies of escalating intensity designed specifically for small hospitals within a vertically integrated healthcare delivery system.

DETAILED DESCRIPTION:
The investigators designed a clustered randomized controlled intervention to evaluate 3 antibiotic stewardship strategies designed for small hospitals. Each hospital was randomized to one of three ASP interventions with increasing levels of intensity and intervention (Programs 1, 2, 3). The investigators felt that clinical equipoise about the effect of ASPs did not exist and randomizing to a no-intervention group was unacceptable. Antibiotic use was compared within each group before and after the intervention. In keeping with other real-world implementation studies, secondary analyses were planned to include an interrupted time series design to evaluate the impact of each strategy. Randomization of hospitals was stratified based on patient volume. Hospital administration and clinical leadership were not blinded to which ASP program they were randomly assigned to, but there were no public announcements. The intervention started March 2014 and ended June 2015.

ELIGIBILITY:
Inclusion Criteria:

* Intermountain Healthcare acute care hospital with < 200 licensed beds
* No formal antibiotic stewardship program in place

Exclusion Criteria:

-All Intermountain Healthcare specialty hospitals, regardless of bed size

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30000 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Total antibiotic use | Total antibiotic use during the 15 months of Intervention (April 1, 2014 through June 30th 2015) was compared to the antibiotic use during the 12 month baseline period (Jan 1 through Dec 31 2013).
  Evaluated change in total antibiotic use between the baseline and intervention periods while accounting for the cluster randomized design.

SECONDARY OUTCOMES:
Broad spectrum antibiotic use | Broad spectrum antibiotic use during the 15 months of Intervention (April 1, 2014 through June 30th 2015) was compared to the broad spectrum antibiotic use during the 12 month baseline period (Jan 1 through Dec 31 2013).
  Evaluated change in broad spectrum antibiotic use between the baseline and intervention periods
Restricted antibiotic use | Restricted antibiotic use during the 15 months of Intervention (April 1, 2014 through June 30th 2015) was compared to the restricted antibiotic use during the 12 month baseline period (Jan 1 through Dec 31 2013).
  Evaluated change in restricted antibiotic use between the baseline and intervention periods
30-day readmission | 30-day readmission rate during the 15 months of Intervention (April 1, 2014 through June 30th 2015) was compared to the 30-day readmission rate during the 12 month baseline period (Jan 1 through Dec 31 2013).
  Evaluated change in 30 day readmission rates between the baseline and intervention periods
30-day mortality | 30-day mortality rate during the 15 months of Intervention (April 1, 2014 through June 30th 2015) was compared to the 30-day mortality rate during the 12 month baseline period (Jan 1 through Dec 31 2013).
  Evaluated change in 30 day mortality rates between the baseline and intervention periods
Hospital length of stay | Average hospital length of stay during the 15 months of Intervention (April 1, 2014 through June 30th 2015) was compared to the average hospital length of stay during the 12 month baseline period (Jan 1 through Dec 31 2013).
  Evaluated change in hospital length of stay between the baseline and intervention periods
Clostridium difficile | C. difficile rate during the 15 months of Intervention (April 1, 2014 through June 30th 2015) was compared to the C. difficile rate during the 12 month baseline period (Jan 1 through Dec 31 2013).
  Evaluated change in Clostridium difficile incidence between the baseline and intervention periods

IPD SHARING:
Plan to Share IPD: No
N/A. No individual patient level data available.

REFERENCES:
- [Background] Stenehjem E, Hersh AL, Sheng X, Jones P, Buckel WR, Lloyd JF, Howe S, Evans RS, Greene T, Pavia AT. Antibiotic Use in Small Community Hospitals. Clin Infect Dis. 2016 Nov 15;63(10):1273-1280. doi: 10.1093/cid/ciw588. Epub 2016 Sep 30. PMID 27694483
- [Derived] Stenehjem E, Hersh AL, Buckel WR, Jones P, Sheng X, Evans RS, Burke JP, Lopansri BK, Srivastava R, Greene T, Pavia AT. Impact of Implementing Antibiotic Stewardship Programs in 15 Small Hospitals: A Cluster-Randomized Intervention. Clin Infect Dis. 2018 Aug 1;67(4):525-532. doi: 10.1093/cid/ciy155. PMID 29790913